CLINICAL TRIAL: NCT06322914
Title: A Novel Scoring System for Predicting the Success of Percutaneous Coronary Interventions in Patients With Chronic Total Occlusion
Brief Title: A Novel Scoring System for Predicting the Success of PCI in Patients With CTO
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Director of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 029
Record Dates: First submitted 2024-03-12; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Chronic Total Occlusion (CTO)
Keywords: Chronic total occlusion (CTO); A Novel Scoring System; the Success of Percutaneous Coronary Interventions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Technical successful group: Technical success of CTO PCI was defined as successful CTO revascularization with achievement of <30% residual diameter stenosis within the treated segment and restoration of antegrade TIMI flow grade 3.
- Technical unsuccessful group: Technical unsuccess of CTO PCI was defined as unsuccessful CTO revascularization（guide wire or stent cannot cross through the lesion）

SUMMARY:
The investigators conducted a retrospective, single-center observational registry upon which one novel scoring system was formed and evaluated for their accuracy in predicting technical success. The investigators reviewed the clinical and angiographic records of 432 patients with 459 CTO lesions who underwent percutaneous recanalization attempts recruited between January 2012 and November 2023. The investigators aims to develop and validate a novel scoring system for predicting CTO-PCI success.

DETAILED DESCRIPTION:
Chronic total occlusions (CTO) accounting for about 15-20% of coronary artery lesions can be challenging and only 10-15% of patients undergo successful percutaneous coronary intervention (PCI) .Thanks to the technological and device advances, the marked improvement of PCI success rates could be seen. However, in contrast to non-CTO lesions, these procedures are accompanied by longer procedure time, contrast and radiation burden, and higher complication rates. The possibility to predict which CTOs are more likely to be treated successfully is still of utmost importance for patient selection. Several scores have been proposed to predict the procedural success rate, such as J-CTO, CL-Score, Progress-Score et al , J-CTO is widely accepted. But Karatasakis et al.showed that these scores performed moderately in predicting technical outcome, while ignoring many factors such as stumpless lesion which may exert an influence on the procedural success. The investigators aims to develop and validate a novel scoring system for predicting CTO-PCI success.

ELIGIBILITY:
Inclusion Criteria:

1. complete occlusion of the coronary artery, confirmed by coronary angiography with TIMI flow grade 0, and occlusion for ≥3 months;
2. presence of angina or angina-equivalent symptoms ; undergo coronary intervention;

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with CTO lesions who underwent percutaneous recanalization attempts recruited between January 2012 and November 2023
Sampling Method: Non-Probability Sample
Enrollment: 493 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2023-11 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
PCI technical success | immediately after PCI
  Technical success of CTO PCI was defined as successful revascularization with <30% residual diameter stenosis and restoration of antegrade TIMI flow grade 3
  of <30% residual diameter stenosis within the treated segment and restoration of antegrade TIMI flow grade 3.

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, Dr,PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Morino Y, Abe M, Morimoto T, Kimura T, Hayashi Y, Muramatsu T, Ochiai M, Noguchi Y, Kato K, Shibata Y, Hiasa Y, Doi O, Yamashita T, Hinohara T, Tanaka H, Mitsudo K; J-CTO Registry Investigators. Predicting successful guidewire crossing through chronic total occlusion of native coronary lesions within 30 minutes: the J-CTO (Multicenter CTO Registry in Japan) score as a difficulty grading and time assessment tool. JACC Cardiovasc Interv. 2011 Feb;4(2):213-21. doi: 10.1016/j.jcin.2010.09.024. PMID 21349461
- [Background] Christopoulos G, Kandzari DE, Yeh RW, Jaffer FA, Karmpaliotis D, Wyman MR, Alaswad K, Lombardi W, Grantham JA, Moses J, Christakopoulos G, Tarar MNJ, Rangan BV, Lembo N, Garcia S, Cipher D, Thompson CA, Banerjee S, Brilakis ES. Development and Validation of a Novel Scoring System for Predicting Technical Success of Chronic Total Occlusion Percutaneous Coronary Interventions: The PROGRESS CTO (Prospective Global Registry for the Study of Chronic Total Occlusion Intervention) Score. JACC Cardiovasc Interv. 2016 Jan 11;9(1):1-9. doi: 10.1016/j.jcin.2015.09.022. PMID 26762904
- [Background] Jin C, Kim MH, Kim SJ, Lee KM, Kim TH, Cho YR, Serebruany VL. Predicting Successful Recanalization in Patients with Native Coronary Chronic Total Occlusion: The Busan CTO Score. Cardiology. 2017;137(2):83-91. doi: 10.1159/000455824. Epub 2017 Feb 8. PMID 28171874
- [Background] Szijgyarto Z, Rampat R, Werner GS, Ho C, Reifart N, Lefevre T, Louvard Y, Avran A, Kambis M, Buettner HJ, Di Mario C, Gershlick A, Escaned J, Sianos G, Galassi A, Garbo R, Goktekin O, Meyer-Gessner M, Lauer B, Elhadad S, Bufe A, Boudou N, Sievert H, Martin-Yuste V, Thuesen L, Erglis A, Christiansen E, Spratt J, Bryniarski L, Clayton T, Hildick-Smith D. Derivation and Validation of a Chronic Total Coronary Occlusion Intervention Procedural Success Score From the 20,000-Patient EuroCTO Registry: The EuroCTO (CASTLE) Score. JACC Cardiovasc Interv. 2019 Feb 25;12(4):335-342. doi: 10.1016/j.jcin.2018.11.020. Epub 2019 Jan 30. PMID 30711551
- [Background] Rigueira J, Aguiar-Ricardo I, Nobre Menezes M, Santos R, Rodrigues T, Cunha N, G Francisco AR, Marques da Costa J, Carrilho Ferreira P, Jorge C, Infante Oliveira E, Duarte J, Torres D, Pinto Cardoso P, Pinto FJ, Canas da Silva P. The CTo-aBCDE score: A new predictor of success in chronic total occlusions. Rev Port Cardiol (Engl Ed). 2020 Oct;39(10):575-582. doi: 10.1016/j.repc.2020.05.007. Epub 2020 Sep 15. English, Portuguese. PMID 32948391